CLINICAL TRIAL: NCT06035796
Title: Performance Study of Targeted Sequencing Technology for Identification of Respiratory Pathogens and Drug Resistance Factor Analysis in VAP Patients
Brief Title: Performance Study of Targeted Sequencing Technology for VAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: Yuting Li111
Record Dates: First submitted 2023-08-25; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-07

CONDITIONS: VAP - Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BALF or sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tNGS(targeted second generation sequencing): tNGS detection of lower respiratory tract samples (BALF) from VAP patients.By means of super-multiple PCR amplification or probe hybridization capture, tNGS can enrich dozens to hundreds of known pathogenic microorganisms and their virulence and drug resistance genes in the samples to be tested, and then conduct high-throughput sequencing.
  Interventions: Device: tNGS
- non-tNGS(non-targeted second generation sequencing): Perform routine clinical testing on lower respiratory tract samples (BALF) from VAP patients and collect patient clinical information. Clinical routine testing includes culture (necessary), microscopy, serology, PCR, etc., and drug sensitivity tests are conducted on positive culture samples as needed.

INTERVENTIONS:
Device: tNGS — By means of super-multiple PCR amplification or probe hybridization capture, tNGS can enrich dozens to hundreds of known pathogenic microorganisms and their virulence and drug resistance genes in the samples to be tested, and then conduct high-throughput sequencing.
  Groups: tNGS(targeted second generation sequencing)

SUMMARY:
Main purpose: To evaluate the feasibility of tNGS for pathogen detection and drug resistance analysis in VAP patients.

Research site and research population:

This study is planned to be conducted in hospitals, targeting VAP patients. Perform clinical routine testing and tNGS testing on lower respiratory tract samples (BALF) from VAP patients, and collect patient clinical information. Clinical routine testing includes culture (necessary), microscopy, serology, PCR, etc., and drug sensitivity tests are conducted on positive culture samples as needed. Finally, compare the consistency of tNGS detection results with clinical culture, comprehensive diagnosis, and drug sensitivity results. Further validation was conducted on consistent negative or inconsistent samples through PCR and mNGS.

DETAILED DESCRIPTION:
The investigators plan to include 150 VAP patients in the ICU. Lower respiratory tract samples (BALF) from VAP patients were routinely tested and tNGS tested, and clinical information was collected. Routine clinical tests include culture (necessary), microscopic examination, serology, PCR, etc., and drug sensitivity tests are performed on positive culture samples as required. Finally, the consistency of tNGS test results with clinical culture, comprehensive diagnosis and drug sensitivity results was compared. The uniformly negative or inconsistent samples were further verified by PCR and mNGS.

ELIGIBILITY:
Inclusion Criteria:

* (1)VAP patients (2) Patients can collect the required test information

Exclusion Criteria:

* (1) Clearly diagnosed as non-infectious patients

  (2) Insufficient samples or patients unwilling to participate

  (3) Life expectancy is less than 24 hours

  (4) Patients' clinical information cannot be obtained

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: VAP patients in the ICU
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
tNGS for pathogen detection rate and drug resistance rate in VAP | 2years
  Evaluating the feasibility of tNGS for pathogen detection rate and drug resistance rate in VAP patients

SECONDARY OUTCOMES:
Consistency rate of pathogen detection of tNGS with clinical practice | 2 years
  1. To compare the consistency rate of TNGs-based pathogen detection with clinical
     culture, multiple clinical detection methods (PCR/ serology, etc.) and comprehensive diagnosis results in the whole and different types of microorganisms (bacteria/viruses/fungi);
  2. To compare the consistency rate of drug resistance results of TNGs-based drug resistance gene test and clinical drug susceptibility test;
  3. To compare the consistency rate of the responsible pathogen based on tNGS semi-quantitative judgment with the clinical comprehensive diagnosis results.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhang, Study Director — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li N, Ma X, Zhou J, Deng J, Gu C, Fei C, Cao L, Zhang Q, Tao F. Clinical application of metagenomic next-generation sequencing technology in the diagnosis and treatment of pulmonary infection pathogens: A prospective single-center study of 138 patients. J Clin Lab Anal. 2022 Jul;36(7):e24498. doi: 10.1002/jcla.24498. Epub 2022 May 27. PMID 35622934
- See also: Clinical application of metagenomic next-generation sequencing technology in the diagnosis and treatment of pulmonary infection pathogens: A prospective single-center study of 138 patients — http://pubmed.ncbi.nlm.nih.gov/35622934/